CLINICAL TRIAL: NCT06896669
Title: Synergistic Effects of Vitamin D and Calcium Supplementation on Hyperglycemia and Dyslipidemia in Patients With Gestational Diabetes
Brief Title: Effects of Vitamin D and Calcium on Hyperglycemia and Dyslipidemia in Patients Gestational Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/24/0848
Record Dates: First submitted 2025-02-20; First posted 2025-03-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Diabetes Mellitus, Gestational
Keywords: Hyperglycemia; Lipid profiles; Pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational; Hyperglycemia | interventions — Cholecalciferol; Calcium

STUDY DESIGN:
Intervention Model Description: It will be randomized control trial, in which intervention group will receive 600 IU of vitamin D3 and 1.5-2 g of calcium daily for 6 weeks and control group will receive a placebo containing no active ingredients.
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm and Interventions (Other): Experimental: Vitamin D3 and calcium This group will be receive vitamin D3 600 IU and 1.5-2 g of calcium. This treatment will be conducted for 6 week per day after meal.
  Interventions: Dietary Supplement: vitamin D3
- Arm and placebo (Other): : This group will receive a placebo containing no active ingredients and it will conducted for 6 weeks per day.
  Interventions: Dietary Supplement: vitamin D3

INTERVENTIONS:
Dietary Supplement: vitamin D3 — 600IU of vitamin D3 and 1.5 to 2g of calcium will be provided for time period of 6 weeks once daily. In addition, Participants dietary intake will be assessed through 24 hours dietary recall.
  Other Names: calcium

SUMMARY:
Gestational diabetes mellitus (GDM) is becoming more common globally as a metabolic disease that occurs during pregnancy and influences the mother and the fetus. It has been linked to preeclampsia, C-section, and a higher lifetime risk of developing type 2 diabetes both for mother and the child. Another complication of GDM is dyslipidemia that also accentuates cardiovascular risks, so the care of lipid profiles is essential for the best pregnancy outcomes. The previous literature review indicates that micronutrients including vitamin D and calcium have a bearing on glucose and lipid profiles. Various studies have established that vitamin D improves the insulin response and lipid profile whereas calcium is vital in insulin and glucose homeostasis. Furthermore, it is revealed that calcium induces vitamin D so that it could undergo its full metabolic effect. Hence, the addition of vitamin D and calcium together may enhance glycemic management and lipid profiles of GDM patients. The aim of the present work is to compare the impact of vitamin D and calcium supplementation on lipid profiles and hyperglycemia in GDM patients. It will measure the major metabolic indices fasting plasma glucose, glycated hemoglobin (HbA1c) and lipid profile (LDL, HDL triglycerides) and review the effect of this on pregnancy outcomes. These outcomes will be assessed by a randomized-controlled trial.

DETAILED DESCRIPTION:
A randomized controlled trial study design will be used to assess the efficacy of vitamin D and calcium supplementation in lipid profiles and glycemic index among women with GDM.

The sample for the study will consist of 60 pregnant women diagnosed with GDM, aged 18-40 years, and between 24-28 weeks of gestation. Recruitment of participants will be done in antenatal clinics linked to [Lady Willingdon Hospital Lahore]. The diagnosis of GDM will be performed according to the results of OGTT following the international criteria.

Participants will be randomly divided to one of two groups:

* Intervention Group: This group will receive 600 IU of vitamin D3 and 1.5-2 g of calcium daily for 6 weeks.
* Control Group: This group will receive a placebo containing no active ingredients.

For randomization, a computer-generated sequence will be used to randomly assign participant into the intervention arm or the placebo arm. The study will be conducted as double blind; the participants and the researchers shall not know the group allocations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women aged 18-40 years.
* Gestational age between 24-28 weeks.
* Diagnosis of GDM based on OGTT results.
* Willingness of participants to provide written informed consent.

Exclusion Criteria:

* Pre-existing diabetes mellitus (type 1 or type 2).
* Chronic kidney or liver disease.
* Use of vitamin D or calcium supplements in the last 3 months.
* Multiple pregnancies (twins, triplets).
* Any major pregnancy complications (e.g., preeclampsia).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Gestational diabetes only occurs during pregnancy, which is female specified only .
Enrollment: 60 (Estimated)
Dates: Start 2025-01-28 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Fasting plasma glucose (FPG) levels | 6 weeks
  fasting plasma glucose measures your blood sugar level post meal after at least 8 hours
HbA1C | 6 weeks
  HbA1C measure glucose level in past 2 to 3 months

SECONDARY OUTCOMES:
lipid profile | 6 weeks
  Lipid profile, including total cholesterol (TC), low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglycerides (TG).

CONTACTS AND LOCATIONS:
Overall Officials: Faryal Gohar, MS, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No